CLINICAL TRIAL: NCT03561870
Title: A Phase II Study of Olaparib in Recurrent IDH-mutant High Grade Gliomas OLAGLI
Brief Title: Olaparib in Recurrent IDH-mutant Glioma
Acronym: OLAGLI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0132; 2018-002584-25 (EudraCT Number)
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2022-04

CONDITIONS: Recurrent IDH; Mutant High Grade Glioma
Keywords: IDH-mutant; recurrent; glioma
MeSH Terms: conditions — Recurrence; Glioma | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental)
  Interventions: Drug: Olaparib 150 MG

INTERVENTIONS:
Drug: Olaparib 150 MG — Olaparaib: 600 mg/day: 300 mg BID (2 x 150 mg tablets taken orally) each 28 days cycle, until disease progression or unacceptable toxicity

SUMMARY:
Recent data demonstrate that in IDH-mutant gliomas, 2 hydroxy-glutarate production induces a homologous recombination defect that renders tumor cells exquisitely sensitive to poly(adenosine 5'-diphosphate-ribose) polymerase (PARP) inhibitors, including olaparib (Lynparza; AstraZeneca). The aim of this open-label phase 2 study is to evaluate the efficacy of olaparib in in recurrent IDH-mutant high grade gliomas based on 6 months progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

1. Affiliation to a French social security system (recipient or assign) excluding AME.
2. Histological confirmation of grade III or IV high-grade glioma or evidence of anaplastic transformation (based on histological or radiological analysis) of a previous grade II glioma
3. Tumor is mutated for IDH1 or IDH2 gene (detected by R132HIDH immunochemistry or IDH1/IDH2 sequencing)
4. Recurrence after radiotherapy and at least one line of alkylating chemotherapy (Temozolomide or PCV (Procarbazine, CCNU, Vincristine) (Surgery at recurrence is allowed before trial inclusion)
5. Recurrence occurring more than 12 weeks from the end of the radiotherapy or occurring outside the irradiated volume
6. Provision of informed consent prior to any study specific procedures
7. Age ≥ 18 years old
8. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:

   Haemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Platelet count ≥ 100 x 109/L total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)) / Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT)) ≤ 2.5 x institutional upper limit of normal

   Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥51 mL/min:

   Estimated creatinine clearance = (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72 a where F=0.85 for females and F=1 for males.
9. KPS ≥ 70
10. Patients must have a life expectancy ≥ 16 weeks.
11. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1.

    Postmenopausal is defined as:

    Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments Luteinizing hormone (LH) and Follicle stimulating hormone (FSH) levels in the post menopausal range for women under 50 radiation-induced oophorectomy with last menses >1 year ago chemotherapy-induced menopause with >1 year interval since last menses surgical sterilisation (bilateral oophorectomy or hysterectomy)
12. Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination [see appendix B for acceptable methods], throughout the period of taking study treatment and for 3 months after last dose of study drug(s) to prevent pregnancy in a partner.
13. Patients is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations.
14. Radiologically measurable disease based on RANO criteria, i. e. at least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by MRI and is suitable for repeated assessment. Tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
15. Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer must be available for central testing. If there is not written confirmation of the availability of an archived tumour sample prior to enrolment the patient is not eligible for the study.
16. For inclusion in the optional biomarker research, patients must fulfil the following criteria:

Provision of informed consent for biomarker research If a patient declines to participate in the optional exploratory genetic research or the optional biomarker research, there will be no penalty or loss of benefit to the patient. The patient will not be excluded from other aspects of the study.

Exclusion Criteria:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
2. Previous enrolment in the present study
3. Participation in another clinical study with an investigational product during the last month
4. Any previous treatment with PARP inhibitor, including olaparib.
5. Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years. Patients with a history of localised triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease.
6. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
7. Patients receiving any systemic chemotherapy or radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
8. Concomitant use of known strong CYP3A inhibitors (eg. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (eg. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks.
9. Concomitant use of known strong (eg. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
10. Persistent toxicities (>Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by previous cancer therapy, excluding alopecia.
11. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
12. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery.
13. Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent.
14. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
15. Breast feeding women.
16. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV).
17. Patients with a known hypersensitivity to olaparib or any of the excipients of the product.
18. Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
19. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
20. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable, for timing refer to inclusion criteria no.8)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
progression free survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: DUCRAY François, PUPH, Study Director — GROUPEMENt Hospitaler EST
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Esparragosa Vazquez I, Sanson M, Chinot OL, Fontanilles M, Rivoirard R, Thomas-Maisonneuve L, Cartalat S, Tabouret E, Appay R, Bonneville-Levard A, Darlix A, Meyronet D, Barritault M, Gueyffier F, Remontet L, Maucort-Boulch D, Honnorat J, Dehais C, Ducray F; POLA Network. Olaparib in recurrent isocitrate dehydrogenase mutant high-grade glioma: A phase 2 multicenter study of the POLA Network. Neurooncol Adv. 2024 May 27;6(1):vdae078. doi: 10.1093/noajnl/vdae078. eCollection 2024 Jan-Dec. PMID 38855053